CLINICAL TRIAL: NCT06424743
Title: Preference of Women With Fibromyalgia Undergoing a Three Different Volumes of Resistance Training: Clinical Trial Randomized Crossover
Brief Title: Preference of Women With Fibromyalgia Undergoing a Three Different Volumes of Resistance Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Marcelo Cardoso de Souza, PT, PhD., Principal Investigator and Professor of Department of Physiotherapy, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UFRNpreference
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Fibromyalgia, Primary; Chronic Pain; Exercise Addiction
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Patients will be allocated to 1 of three groups: 1 set, 2 sets, or 3 sets of resistance exercise. In the next sessions they will be allocated to the series he has not performed yet.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 set (Experimental): Training A Bench press, Pull front, Leg press and seated flexor
  1 series 10 repetitions with 60% 1RM, 2' minute interval
  Interventions: Other: exercise
- 2 sets (Experimental): Training B Bench press, Pull front, Leg press and seated flexor 2 series 10 repetitions with 60% 1RM, 2' minute interval
  Interventions: Other: exercise
- 3 sets (Experimental): Training C Bench press, Pull front, Leg press and seated flexor 3 series 10 repetitions with 60% 1RM, 2' minute interval
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — exercise programs with different volumes
  Other Names: resistance exercises

SUMMARY:
Fibromyalgia is a painful syndrome of unknown etiology, which affects 2% of world population, with symptoms such as: pain, unrefreshing sleep, fatigue and mood disorders. It is already established in the literature that resistance training is part of the non- pharmacological treatment for patients with fibromyalgia. The big gap is about the quantity adequate and/or recommended exercise volume, despite some studies with exercise volumes different resistance trainings show improvements, we do not have a direction, besides We still do not know whether there is a preference for these patients in different resistance training volumes.

DETAILED DESCRIPTION:
Objective: Assess training volume preference resisted in women with fibromyalgia.

Method: Crossover randomized clinical trial, randomized and blind. 36 women with fibromyalgia will be evaluated, who will undergo three resistance training programs with different training volumes. The primary outcome will be patient preference in relation to training volumes, and the secondary ones will be the patient expectation, pain intensity, affect and subjective perception of exertion.

Analysis statistics: For the primary outcome preference, the number of choices will be counted of the 3 types of training in percentage form. Regarding the analysis of the primary outcome we will summarize the patient's preference in a contingency table, we will compare the proportions using the Chi-square test, and finally we will check the effect size of the observed differences. For secondary outcomes, statistical analyzes will be performed by a blind statistician using commercial software. The Kolmogorov-Smirnov test will be applied to verify the distribution of data and Levene's test will be used to analyze the homogeneity of variance. The Bonferroni test will be used in post hoc analyzes to determine whether there are differences between the groups at different intervention times. One 5% significance level and 95% CI will be adopted for all statistical analyses. ethic and dissemination: The results of the study will be disseminated to participants and subjected to a peer-reviewed journal and scientific meetings.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 65
* Have a diagnosis of fibromyalgia according to the ACR 2016 criteria

Exclusion Criteria:

* Have performed resistance training in the last 6 months
* Having another associated rheumatic condition
* Have a trip or appointment scheduled that requires absence for the next 4 (four) weeks from the start of the survey;
* Women with musculoskeletal injuries in the upper and/or lower limbs
* Have heart problems that prevent maximal efforts and submaximums

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Choose one of the workouts according to your preference | 28 day
  Preference will be assessed through the following question: "After carrying out the training sessions, which one did you prefer? Why?".

SECONDARY OUTCOMES:
Change in Expectation | baseline
  The Likert Scale will be used for expectations in relation to treatment. That scale aims to assess the participant's expectations at the beginning of the study in relation to the treatment they will receive with the following questions: • "Do you think that by starting the training session with 1 set, you will: (1) get much worse, (2) get a little worse, (3) neither get better nor get worse (4) get better little and (5) improve a lot".
  * "Do you think that by starting the training session with 2 sets, you will: (1) get much worse, (2) get a little worse, (3) neither get better nor get worse (4) get better little and (5) improve a lot".
  * "Do you think that by starting the training session with 3 sets, you will: (1) get much worse, (2) get a little worse, (3) neither get better nor get worse (4) get better little and (5) improve a lot".
Change in Pain intensity | baseline, 28 day
  Generalized pain intensity will be assessed using the Numerical Pain Scale (END), a self-report instrument validated for Portuguese. END has a sequence of numbers (from 0 to 10), where 0 represents "no pain" and 10 represents "the worst pain that you can imagine."
Change in Affection | baseline, 28 day
  Affect scale will monitor pleasure or displeasure during the three resistance training will be carried out through the application of the affective valence scale (VA).
  The scale is quantified as follows: +5 to -5, corresponding, respectively, to the two antagonistic descriptors of feelings during physical exercise and/or physical activity, which may be: "very good" and "very bad".
Change in Subjective perception of exertion | baseline, 28 day
  The quantification of the intensity of each resistance training session will be determined using the session's subjective perception of exertion (RPE) method
  . To this end, the following question: "How was your training session?" The answer will be provided, as recommended, 30 min after the end of the session, based on an adapted Borg scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Marcelo Cardoso de Souza, Natal, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No
there is not a plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Result] Silva HJA, Assuncao Junior JC, de Oliveira FS, Oliveira JMP, Figueiredo Dantas GA, Lins CAA, de Souza MC. Sophrology versus resistance training for treatment of women with fibromyalgia: A randomized controlled trial. J Bodyw Mov Ther. 2019 Apr;23(2):382-389. doi: 10.1016/j.jbmt.2018.02.005. Epub 2018 Feb 12. PMID 31103124
- [Derived] Cavalcanti BH, Pontes-Silva A, Souza CG, Avila MA, de Souza MC. Do Fibromyalgia Patients Have a Preferred Resistance Training Volume? Protocol for a Randomized Crossover Clinical Trial. Physiother Res Int. 2025 Oct;30(4):e70101. doi: 10.1002/pri.70101. PMID 40886126